CLINICAL TRIAL: NCT01244581
Title: Oral Amoxicillin-clavulanate in Treating Acute Otitis Media in Children: Randomized Double-blind Placebo-controlled Study Including Daily Monitoring With Tympanometry
Brief Title: Amoxicillin-clavulanate in Treating Acute Otitis Media Evaluated by Daily Tympanometry
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Terhi Tapiainen, M.D., Ph.D., University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OYS_Tapiainen_001
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Otitis Media, Suppurative
Keywords: middle ear effusion; amoxicillin-clavulanate; tympanometry
MeSH Terms: conditions — Otitis Media, Suppurative; Otitis Media with Effusion | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin-clavulanate (Experimental): Oral amoxicillin-clavulanate 40 mg/kg/day divided in two daily doses for 7 days
  Interventions: Drug: Amoxicillin-clavulanate
- Placebo (Placebo Comparator)
  Interventions: Drug: Amoxicillin-clavulanate; Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin-clavulanate — Amoxicillin-clavulanate 40 mg/kg/day in two daily doses for 7 days
  Other Names: Clavurion
Drug: Placebo — Placebo mixture in two daily doses for 7 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy of amoxicillin-clavulanate in treating acute otitis media in children. The primary end point is time to disappearance of middle ear effusion which monitored by daily tympanometry performed by families and study physicians.

ELIGIBILITY:
Inclusion Criteria:

* Children with acute otitis media

Exclusion Criteria:

* Amoxicillin allergy
* Tympanic membrane perforation
* Tympanostomy tubes (current)
* Complication of acute otitis media such as mastoiditis

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 1999-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Time (days) to disappearance of middle ear effusion | Within 60 days
  Disappearance of middle ear effusion is defined as the first day of receiving a normal tympanogram (A-curve) in tympanometry.

SECONDARY OUTCOMES:
Time (days) to disappearance of pain | Within 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Matti Uhari, Professor, Study Director — University of Oulu; Terhi Tapiainen, MD, PhD, Principal Investigator — University of Oulu
Locations (2):
- Finland (2):
  - Department of Pediatrics, Oulu University Hospital, Oulu
  - Lääkärikeskus Mehiläinen, Oulu

REFERENCES:
- [Derived] Tapiainen T, Kujala T, Renko M, Koivunen P, Kontiokari T, Kristo A, Pokka T, Alho OP, Uhari M. Effect of antimicrobial treatment of acute otitis media on the daily disappearance of middle ear effusion: a placebo-controlled trial. JAMA Pediatr. 2014 Jul;168(7):635-41. doi: 10.1001/jamapediatrics.2013.5311. PMID 24797294